CLINICAL TRIAL: NCT05410093
Title: Clinical Efficacy Analysis of Resveratrol in the Treatment of Primary Ovarian Insufficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: LCYJ-B05
Record Dates: First submitted 2022-05-16; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-02

CONDITIONS: Primary Ovarian Insufficiency
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Resveratrol; Vitamin E; Tocopherols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients who taking Resveratrol (Experimental): Take RES (250mg, NuMedica, FDA approved) at a dose of 250mg per day for three months
  Interventions: Drug: Resveratrol
- Patients who taking VitE (Active Comparator): Take vitamin E at a dose of 100 mg per day for three months
  Interventions: Drug: Vitamin E

INTERVENTIONS:
Drug: Resveratrol — Take Resveratrol (250mg, NuMedica, FDA approved) at a dose of 250mg per day for three months
  Other Names: Res
  Arms: Patients who taking Resveratrol
Drug: Vitamin E — Take vitamin E at a dose of 100 mg per day for three months
  Other Names: tocopherol
  Arms: Patients who taking VitE

SUMMARY:
Resveratrol is a natural plant antitoxin widely found in grapes, mulberries, and other plants. Resveratrol mediates a variety of pharmacological effects, including antioxidant, immunomodulatory, anti-inflammatory, and anti-apoptotic, and plays a protective and therapeutic role in the development of several ROS-related diseases, including POI/POF.

DETAILED DESCRIPTION:
The preliminary experiments of the investigators' group examined the gene expression in ovarian granulosa cells of POI patients and normal controls using high-throughput sequencing technology. The investigators found that the expression of NOX complex NCF1, NCF2, NCF4 and CYBB subunit genes were upregulated in ovarian granulosa cells of POI patients compared with normal controls, suggesting that the development of POI may be related to the NOX complex subunit gene and The development of POI may be related to the abnormal expression of genes and proteins of NOX complex subunits. Based on the results of previous experiments and available literature reports, investigators compared ovarian function, embryonic laboratory indices, pregnancy outcome and cellular level NOX/ROS/oxidative stress changes of POI patients in the RES-treated and non-RES-treated groups by collecting blood and ovarian granulosa cell samples to analyze the effects, mechanisms of action and specific RES application in antioxidant therapy for POI NOX subunit targets to provide a reliable scientific basis for the clinical treatment of POI by RES.

ELIGIBILITY:
Inclusion Criteria:

1. Amenorrhea or oligomenorrhea at least 4 months and two (>4 weeks interval) basal FSH≥10mIU/ml；
2. The women aged <40 years old；
3. Informed consent, voluntary experiment.

Exclusion Criteria:

1. Pregnant and lactating patients;
2. Patients with endometriosis, adenomyosis, endometrial lesions (submucosal fibroids, endometrial polyps, etc.), uterine fibroids>4 cm or hysterectomy;
3. Patients with adrenal cortical hyperplasia or tumour；
4. Ovarian neoplasms patients；
5. Hydrosalpinx patients；
6. Hyperprolactinemia patients；
7. Patients who are participating in other clinical trials or have participated in other clinical trials within the past three months;
8. Patients with a suspected or real history of alcohol and drug abuse;
9. Known allergy to the investigational drug or its components;
10. Other patients were deemed unsuitable for participation in this trial by the investigator.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Follicle-stimulating hormone (FSH) | Third day of menstruation
  Compare Differences
Luteinizing hormone (LH) | Third day of menstruation
  Compare Differences

SECONDARY OUTCOMES:
Anti-Mullerian hormone (AMH) | Third day of menstruation
  Compare Differences
Estradiol hormone (E2) | Third day of menstruation
  Compare Differences
Testosterone (T) | Third day of menstruation
  Compare Differences

CONTACTS AND LOCATIONS:
Overall Officials: wang xia, Master, Study Chair — Hospital affiliated of nantong university
Locations (1):
- B ultrasound, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT05410093/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT05410093/SAP_001.pdf